CLINICAL TRIAL: NCT05784844
Title: Antimicrobial Revision in Patients With Persistent Febrile Neutropenia: A Prospective, Randomized Trial
Brief Title: Antimicrobial Revision in Persistent Febrile Neutropenia
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was never initiated or activated - Reason was lack of funding
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00088805
Record Dates: First submitted 2023-03-02; First posted 2023-03-27 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-02

CONDITIONS: Febrile Neutropenia
Keywords: acute myeloid leukemia; acute lymphocytic leukemia
MeSH Terms: conditions — Febrile Neutropenia; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Meropenem; Micafungin

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, open-label, single center trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Meropenem Arm (Active Comparator): Patients who meet inclusion criteria may be randomized to meropenem (routine standard of care) dose according to local dosing guidelines to include the use of extended-infusions and adjustments to account for renal function. Duration will be managed by the primary team.
  Interventions: Drug: Meropenem
- Micafungin Arm (Active Comparator): Patients who meet inclusion criteria may be randomized to micafungin dosed as 150mg intravenously every 24 hours according to local dosing guidelines. Duration will be managed by the primary team.
  Interventions: Drug: Micafungin

INTERVENTIONS:
Drug: Meropenem — Carbapenem antibiotic
  Other Names: Merrem
  Arms: Meropenem Arm
Drug: Micafungin — Echinocandin antifungal
  Other Names: Mycamine
  Arms: Micafungin Arm

SUMMARY:
Febrile neutropenia is often seen in patients with hematologic malignancies who receive cytotoxic chemotherapy. These patients are usually placed on posaconazole prophylaxis upon starting chemotherapy. If an episode of febrile neutropenia occurs, generally an anti-pseudomonal beta lactam, like cefepime or piperacillin-tazobactam, is initiated. In patients who continue to fever on these agents, the optimal method of antimicrobial revision has yet to be determined.

DETAILED DESCRIPTION:
In this prospective, randomized, open-label, single-center trial, the primary objective is to compare the clinical efficacy of two approaches to antimicrobial revision among patients with persistent febrile neutropenia. Neutropenic patients on cefepime or piperacillin-tazobactam who continue to fever for greater than 96 hours will be randomized to receive either meropenem or micafungin dosed according to local guidelines. The primary outcome is a global success rate including a composite of defervescence within 72 hours of meropenem or micafungin initiation, absence of signs or symptoms of infection, and no modification to antimicrobial regimen after initiation of meropenem or micafungin. The secondary outcomes to be collected include in-hospital mortality or discharge to hospice, hospital length of stay, time to defervescence, days of therapy of meropenem or micafungin, rate of Clostridioides difficile infection on meropenem or micafungin, and cause of any proven breakthrough infection while on meropenem or micafungin.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Diagnosis of hematologic malignancy
* Receiving chemotherapy as treatment of hematologic malignancy
* Neutropenia defined as an absolute neutrophil count (ANC) ≤ 500 cells/mm3 or an ANC ≤ 1000 cells/mm3 with a predicted decline to < 500 cells/mm3 within 48 hours
* Prescribed cefepime or piperacillin-tazobactam as initial treatment for febrile neutropenia
* Persistent fever for ≥ 96 hours since initiation of cefepime or piperacillin-tazobactam OR recurrent fever that occurs ≥ 96 hours since initiation of cefepime or piperacillin-tazobactam (fever defined as single temperature of ≥ 38.3°C (101°F) or a temperature of ≥ 38°C (100.4°F) on two consecutive measures separated by at least one hour)
* Receipt of posaconazole as neutropenia prophylaxis for at least 3 calendar days

Exclusion Criteria:

* Clinically or microbiologically confirmed infection at time of enrollment, For example, a positive culture or rapid diagnostic test, positive imaging (X-ray, CT, MRI) or biomarker, such as galactomannan, that is consistent with infection
* History of infection with organism known to be resistant to meropenem or micafungin
* Documented allergy to carbapenems or echinocandins
* Concomitant use of valproic acid
* Uncontrolled seizure disorder
* Pregnancy
* Previous enrollment in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Global Success Rate | Hour 72
  Percentage of study candidates who meet all of the following criteria:
  * Defervescence, as defined by a temperature < 38°C (100.4°F) sustained for at least 24 consecutive hours, within 72 hours of meropenem or micafungin initiation
  * Absence of signs or symptoms of infection within 72 hours of meropenem or micafungin initiation including but not limited to hypotension, erythema at catheter sites or cellulitis, positive imaging concerning for infection (e.g., pneumonia, osteomyelitis, abscesses etc.), positive cultures or rapid diagnostic tests, positive biomarkers (e.g. galactomannan), dysuria, hypothermia (≤ 35°C or ≤ 95°F) etc.
  * No modification to antimicrobial regimen after initiation of meropenem or micafungin unless the antibiotic modification is considered de-escalation (e.g. discontinuation of vancomycin)

SECONDARY OUTCOMES:
Number of Subjects In-hospital mortality or discharge to hospice | From hospital admission to death/discharge to hospice, up to 4 days
  Death during in-hospital admission or discharge from in-hospital admission to hospice care
Hospital length of stay (days) | From hospital admission to discharge, up to 4 days
  Number of days admitted to hospital
Time to defervescence (hours) | through study completion, an average of 4 days
  * Time of defervescence defined as the beginning of the 24 consecutive hour afebrile period
  * Time to defervescence defined as the time in hours from the initial documented fever to the beginning of the 24 consecutive hour afebrile period
Days of therapy of meropenem or micafungin | through study completion, an average of 4 days
  1 antibiotic x the number of days administered, any calendar day in which at least one dose is given counts as a full day of therapy - Time in days from initiation to discontinuation of meropenem or micafungin
Rate of Clostridioides difficile infection on meropenem or micafungin | through study completion, an average of 4 days
  Percentage of patients who develop Clostridioides difficile infection while on meropenem or micafungin
Collection of Causes of any proven breakthrough infection while on meropenem or micafungin | through study completion, an average of 4 days
  Collection of origin of proven breakthrough infection

CONTACTS AND LOCATIONS:
Overall Officials: John Williamson, PharmD, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] National Comprehensive Cancer Network (NCCN) Clinical Practice Guidelines in Oncology (NCCN Guidelines®). Prevention and Treatment of Cancer-Related Infections Version 1.2022. Accessed July 12, 2022. https://www.nccn.org/guidelines/guidelines-detail?category=3&id=1457
- [Background] Freifeld AG, Bow EJ, Sepkowitz KA, Boeckh MJ, Ito JI, Mullen CA, Raad II, Rolston KV, Young JA, Wingard JR; Infectious Diseases Society of America. Clinical practice guideline for the use of antimicrobial agents in neutropenic patients with cancer: 2010 update by the infectious diseases society of america. Clin Infect Dis. 2011 Feb 15;52(4):e56-93. doi: 10.1093/cid/cir073. PMID 21258094
- [Background] Averbuch D, Orasch C, Cordonnier C, Livermore DM, Mikulska M, Viscoli C, Gyssens IC, Kern WV, Klyasova G, Marchetti O, Engelhard D, Akova M; ECIL4, a joint venture of EBMT, EORTC, ICHS, ESGICH/ESCMID and ELN. European guidelines for empirical antibacterial therapy for febrile neutropenic patients in the era of growing resistance: summary of the 2011 4th European Conference on Infections in Leukemia. Haematologica. 2013 Dec;98(12):1826-35. doi: 10.3324/haematol.2013.091025. PMID 24323983
- [Background] Zimmer AJ, Freifeld AG. Optimal Management of Neutropenic Fever in Patients With Cancer. J Oncol Pract. 2019 Jan;15(1):19-24. doi: 10.1200/JOP.18.00269. PMID 30629902
- [Background] Walsh TJ, Teppler H, Donowitz GR, Maertens JA, Baden LR, Dmoszynska A, Cornely OA, Bourque MR, Lupinacci RJ, Sable CA, dePauw BE. Caspofungin versus liposomal amphotericin B for empirical antifungal therapy in patients with persistent fever and neutropenia. N Engl J Med. 2004 Sep 30;351(14):1391-402. doi: 10.1056/NEJMoa040446. PMID 15459300
- [Background] Oyake T, Kowata S, Murai K, Ito S, Akagi T, Kubo K, Sawada K, Ishida Y. Comparison of micafungin and voriconazole as empirical antifungal therapies in febrile neutropenic patients with hematological disorders: a randomized controlled trial. Eur J Haematol. 2016 Jun;96(6):602-9. doi: 10.1111/ejh.12641. Epub 2015 Aug 26. PMID 26216048
- [Background] Oztoprak N, Piskin N, Aydemir H, Celebi G, Akduman D, Keskin AS, Gokmen A, Engin H, Ankarali H. Piperacillin-tazobactam versus carbapenem therapy with and without amikacin as empirical treatment of febrile neutropenia in cancer patients: results of an open randomized trial at a university hospital. Jpn J Clin Oncol. 2010 Aug;40(8):761-7. doi: 10.1093/jjco/hyq046. Epub 2010 Apr 28. PMID 20427546
- [Background] Wang Y, Du Z, Chen Y, Liu Y, Yang Z. Meta-analysis: combination of meropenem vs ceftazidime and amikacin for empirical treatment of cancer patients with febrile neutropenia. Medicine (Baltimore). 2021 Feb 26;100(8):e24883. doi: 10.1097/MD.0000000000024883. PMID 33663117
- [Background] Nakane T, Tamura K, Hino M, Tamaki T, Yoshida I, Fukushima T, Tatsumi Y, Nakagawa Y, Hatanaka K, Takahashi T, Akiyama N, Tanimoto M, Ohyashiki K, Urabe A, Masaoka T, Kanamaru A; Japan Febrile Neutropenia Study Group. Cefozopran, meropenem, or imipenem-cilastatin compared with cefepime as empirical therapy in febrile neutropenic adult patients: A multicenter prospective randomized trial. J Infect Chemother. 2015 Jan;21(1):16-22. doi: 10.1016/j.jiac.2014.08.026. Epub 2014 Sep 17. PMID 25239059
- [Background] Nakagawa Y, Suzuki K, Ohta K, Hino M, Ohyashiki K, Kanamaru A, Tamura K, Urabe A, Masaoka T; Japan Febrile Neutropenia Study Group. Prospective randomized study of cefepime, panipenem, or meropenem monotherapy for patients with hematological disorders and febrile neutropenia. J Infect Chemother. 2013 Feb;19(1):103-11. doi: 10.1007/s10156-012-0466-8. Epub 2012 Sep 5. PMID 22948387
- [Background] Ratliff CM, Beardsley JR, Kennedy L, Ohl C, Johnson JW, Luther VP, William JC. Efficacy of doripenem compared with meropenem for treatment of febrile neutropenia among patients who became febrile while on cefepime or piperacillin-tazobactam. Poster Presented at: Infectious Diseases Society of America Annual Meeting; October 21, 2011; Boston, MA. https://idsa.confex.com/idsa/2011/webprogram/Paper30902.html
- See also: National Comprehensive Cancer Network (NCCN) Clinical Practice Guidelines in Oncology (NCCN Guidelines®) — https://www.nccn.org/guidelines/guidelines-detail?category=3&id=1457